CLINICAL TRIAL: NCT03053427
Title: Gabapentin Enacarbil Post-marketing Clinical Study A Randomized, Double-blind, Placebo-controlled, Parallel-group Study in Subjects With Restless Legs Syndrome.
Brief Title: A Study of Oral Dosing of Gabapentin Enacarbil in Japanese Restless Legs Syndrome Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8825-CL-0101
Record Dates: First submitted 2017-02-12; First posted 2017-02-15 (Actual); Results first posted 2019-07-10 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Restless Legs Syndrome (RLS)
Keywords: Restless Legs Syndrome; ASP8825; Gabapentin enacarbil
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo was administered orally once daily after the evening meal.
  Interventions: Drug: Placebo
- Gabapentin enacarbil (Experimental): Gabapentin enacarbil was administered orally once daily after the evening meal. Participants with an estimated creatinine clearance of ≥ 60 mL/min to < 90 mL/min at the start of the run-in period were administrated gabapentin enacarbil 300 mg for 1 week followed by gabapentin enacarbil 600 mg for 11 weeks.
  Interventions: Drug: Gabapentin enacarbil

INTERVENTIONS:
Drug: Placebo — Oral administration
  Arms: Placebo
Drug: Gabapentin enacarbil — Oral administration
  Other Names: Regnite
  Arms: Gabapentin enacarbil

SUMMARY:
The objective of this study was to assess the efficacy of once-daily oral administration of gabapentin enacarbil versus placebo, based on the change in International Restless Legs Syndrome Rating Scale (IRLS) score in participants with moderate-to-severe idiopathic restless legs syndrome. This study also assessed the safety of Gabapentin enacarbil.

DETAILED DESCRIPTION:
After 1 week run in period with single-blind placebo, participants meeting the inclusion and none of the exclusion criteria were randomized to receive double-blind treatment with either gabapentin enacarbil 600 mg or placebo for 12 weeks treatment period. After then, single-blind placebo was given for 1 week for follow-up observation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Restless Legs Syndrome (RLS), based on the International Restless Legs Syndrome Study Group (IRLSSG) Diagnostic Criteria.
* Subject has reported history of RLS symptoms for at least 15 days in the month prior to the first dosing; if on treatment, this frequency of symptoms was started before treatment.
* Subject with International Restless Legs Syndrome Rating Scale (IRLS) score ≥ 15.
* Subject has discontinued dopamine agonists, and/or gabapentin at least 1 week prior to the first dosing.
* Subject has discontinued other treatments for RLS at least 2 weeks prior to the first dosing.
* Female subject must either:

Be of non-childbearing potential:

* Post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
* documented surgically sterile

Or, if of childbearing potential:

* Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
* And have a negative urine pregnancy test at Screening
* And, if heterosexually active, agree to consistently use two forms of highly effective birth control starting at Screening and throughout the study period and for 28 days after the final study drug administration.

  * Female subject must agree not to breastfeed starting at Screening and throughout the study period, and for 28 days after the final study drug administration.
  * Female subject must not donate ova starting at Screening and throughout the study period, and for 28 days after the final study drug administration.
  * Subject agrees not to participate in another interventional study while on treatment.
  * Subject with a Body Mass Index of ≥ 18.5 and < 30.
  * Subject with estimated creatinine clearance of ≥ 60 mL/min.

Exclusion Criteria:

* Subject has a sleep disorder that may significantly affect the assessment of RLS.
* Subject has a history of RLS symptom augmentation or end-of-dose rebound with previous dopamine agonist treatment.
* Subject has neurologic disease or movement disorder.
* Subject has poorly controlled diabetes, iron deficiency anemia, or are currently taking any sedative/hypnotic.
* Subject has a history of suicide attempt within 6 months prior to informed consent.
* Subject has a high level of Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST).
* Subject is currently suffering from moderate or severe depression.
* Subject has a history of alcohol dependence or drug abuse, or subject had alcohol or drug abuse or dependence in the last 1 year.
* Subject is a shift worker, professional driver, or operator of dangerous machinery.
* Subject has clinically significant or unstable medical conditions.
* Subject has a history of hypersensitivity reaction to gabapentin.
* Subject has previously taken pregabalin, gabapentin enacarbil, or the study drug of Gabapentin enacarbil.
* Subject has participated in a clinical study for another investigational drug or medical device or post-marketing clinical study within 12 weeks (84 days) prior to the first dosing, or is currently participating in any of these studies.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (46):
- Japan (46):
  - Site JP00025, Nagoya, Aichi-ken
  - Site JP00029, Nagoya, Aichi-ken
  - Site JP00040, Nagoya, Aichi-ken
  - Site JP00006, Kitakyushu, Fukuoka
  - Site JP00022, Kitakyushu, Fukuoka
  - Site JP00002, Sapporo, Hokkaido
  - Site JP00003, Sapporo, Hokkaido
  - Site JP00004, Sapporo, Hokkaido
  - Site JP00023, Sapporo, Hokkaido
  - Site JP00041, Kawanishi, Hyōgo
  - Site JP00005, Kobe, Hyōgo
  - Site JP00038, Kawasaki, Kanagawa
  - Site JP00007, Yokohama, Kanagawa
  - Site JP00017, Yokohama, Kanagawa
  - Site JP00049, Yokohama, Kanagawa
  - Site JP00050, Yokohama, Kanagawa
  - Site JP00009, Yokosuka, Kanagawa
  - Site JP00032, Sakai, Osaka
  - Site JP00043, Tokorozawa, Saitama
  - Site JP00012, Arakawa City, Tokyo
  - Site JP00001, Chōfu, Tokyo
  - Site JP00028, Chōfu, Tokyo
  - Site JP00018, Chūō, Tokyo
  - Site JP00024, Chūō, Tokyo
  - Site JP00048, Meguro City, Tokyo
  - Site JP00034, Musashino, Tokyo
  - Site JP00046, Nakano City, Tokyo
  - Site JP00019, Ōta-ku, Tokyo
  - Site JP00011, Shibuya City, Tokyo
  - Site JP00013, Shinagawa, Tokyo
  - Site JP00015, Shinagawa, Tokyo
  - Site JP00016, Shinagawa, Tokyo
  - Site JP00008, Shinjuku, Tokyo
  - Site JP00014, Shinjuku, Tokyo
  - Site JP00021, Shinjuku, Tokyo
  - Site JP00031, Chiba
  - Site JP00036, Fukuoka
  - Site JP00020, Kyoto
  - Site JP00035, Kyoto
  - Site JP00010, Osaka
  - Site JP00026, Osaka
  - Site JP00037, Osaka
  - Site JP00039, Osaka
  - Site JP00047, Osaka
  - Site JP00030, Saitama
  - Site JP00044, Saitama

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderate to severe idiopathic restless legs syndrome were enrolled in 51 study sites in Japan.
Pre-assignment Details: Participants received single-blind placebo for 1 week (run-in period). Subsequently, eligible participants were randomized to receive gabapentin enacarbil or placebo orally once daily after dinner for 12 weeks (treatment period).
Groups:
- Gabapentin Enacarbil: Gabapentin enacarbil was administered orally once daily after the evening meal. Participants with an estimated creatinine clearance of ≥ 60 mL/min to < 90 mL/min at the start of the run-in period were administrated gabapentin enacarbil 300 mg for 1 week (upward titration period) followed by gabapentin enacarbil 600 mg for 11 weeks.
Period: Overall Study
Arm/Group | Placebo | Gabapentin Enacarbil
Started | 186 | 189
Completed | 173 | 173
Not Completed | 13 | 16
Not completed — Adverse Event | 4 | 4
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Worsening of the target disease | 0 | 1
Not completed — Protocol Deviation | 3 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Miscellaneous | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) consisted of all participants given at least one dose of the study drug for the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gabapentin Enacarbil | Total
Number analyzed (Participants) | 186 | 189 | 375
Age, Continuous [Mean (Standard Deviation); unit: year] | 52.2 (12.4) | 51.1 (13.5) | 51.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 90 | 169
  Male | 107 | 99 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 186 | 189 | 375
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 186 | 189 | 375
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
International Restless Legs Syndrome Rating Scale (IRLS) score [Mean (Standard Deviation); unit: units on a scale] — The IRLS consisted of 10-item scale for assessing severity of restless legs syndrome with each item ranging from 0 (no symptoms) to 4 (very severe symptoms). The total IRLS score ranges from 0 to 40. Higher IRLS score indicated greater disease activity. Population: Data were provided for the full analysis set (FAS), which included all participants who received study drug and were evaluated for at least one efficacy (either primary or secondary) endpoint during the treatment period.
  units on a scale
    number analyzed (Participants) | 186 | 188 | 374
    (all) | 23.8 (5.4) | 23.7 (5.2) | 23.7 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Restless Legs Syndrome Rating Scale (IRLS) Score at Week 12
Description: The IRLS consisted of 10-item scale for assessing severity of restless legs syndrome (RLS) with each item ranging from 0 (no symptoms) to 4 (very severe symptoms). The total IRLS score ranges from 0 to 40. Higher IRLS score indicated greater disease activity. Mixed Model of Repeated Measurements (MMRM) model with compound symmetry as a covariance structure was used. The explanatory variables of the model included treatment group, IRLS score at baseline, age category, estimated creatinine clearance category, time point, and interaction of treatment group and time point.
Time Frame: Baseline and week 12
Population: Full Analysis Set (FAS) consisted of all participants who received the study drug for the treatment period and were evaluated for at least one efficacy (either primary or secondary) endpoint during the treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 188
units on a scale | -10.5 [-11.4 to -9.5] | -11.7 [-12.6 to -10.7]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin Enacarbil; MMRM with compound symmetry as the covariance structure was used. The explanatory variables of the model included treatment group, IRLS score at baseline, age category, estimated creatinine clearance category, time point, and interaction of treatment group and time point; Test type: Superiority; p = 0.088, Mixed Model of Repeated Measurements; LSM difference = -1.2, 95% CI 2-sided [-2.6 to 0.2], Standard Error of Mean 0.7

2. Secondary Outcome: Change From Baseline in IRLS Score at Each Time Point
Description: ANCOVA model with the baseline value as a covariate was used.
Time Frame: Baseline and weeks 1, 2, 4, 6, 8, 10, 12 and EoT (week 12)
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 188
units on a scale
  Week 1: number analyzed (Participants) | 186 | 186
  Week 1 | -3.1 [-3.9 to -2.3] | -4.2 [-5.0 to -3.4]
  Week 2: number analyzed (Participants) | 181 | 184
  Week 2 | -4.3 [-5.2 to -3.4] | -5.8 [-6.7 to -4.9]
  Week 4: number analyzed (Participants) | 182 | 180
  Week 4 | -6.0 [-6.9 to -5.0] | -7.5 [-8.4 to -6.5]
  Week 6: number analyzed (Participants) | 180 | 176
  Week 6 | -7.4 [-8.4 to -6.3] | -8.8 [-9.9 to -7.8]
  Week 8: number analyzed (Participants) | 177 | 174
  Week 8 | -8.8 [-9.8 to -7.8] | -9.8 [-10.8 to -8.8]
  Week 10: number analyzed (Participants) | 177 | 173
  Week 10 | -9.6 [-10.6 to -8.5] | -11.2 [-12.3 to -10.2]
  Week 12: number analyzed (Participants) | 174 | 173
  Week 12 | -10.5 [-11.6 to -9.4] | -11.9 [-13.0 to -10.8]
  EoT | -10.2 [-11.4 to -9.1] | -11.1 [-12.2 to -9.9]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin Enacarbil; LMS difference (gabapentin enacarbil group minus placebo group) of the changes in IRLS score from baseline was calculated by visit, using ANCOVA model with the baseline value as a covariate; Test type: Superiority; p = 0.051, ANCOVA; Time frame: week 1; LSM difference = -1.1, 95% CI 2-sided [-2.2 to 0.0], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Placebo vs Gabapentin Enacarbil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.020, ANCOVA; Time frame: week 2; LSM difference = -1.5, 95% CI 2-sided [-2.8 to -0.2], Standard Error of Mean 0.7
Statistical Analysis 3: Comparison: Placebo vs Gabapentin Enacarbil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.028, ANCOVA; Time frame: week 4; LSM difference = -1.5, 95% CI 2-sided [-2.9 to -0.2], Standard Error of Mean 0.7
Statistical Analysis 4: Comparison: Placebo vs Gabapentin Enacarbil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.043, ANCOVA; Time frame: week 6; LSM difference = -1.5, 95% CI 2-sided [-2.9 to -0.0], Standard Error of Mean 0.7
Statistical Analysis 5: Comparison: Placebo vs Gabapentin Enacarbil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.184, ANCOVA; Time frame: week 8; LSM difference = -1.0, 95% CI 2-sided [-2.4 to 0.5], Standard Error of Mean 0.7
Statistical Analysis 6: Comparison: Placebo vs Gabapentin Enacarbil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.027, ANCOVA; Time frame: week 10; LSM difference = -1.7, 95% CI 2-sided [-3.1 to -0.2], Standard Error of Mean 0.7
Statistical Analysis 7: Comparison: Placebo vs Gabapentin Enacarbil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.087, ANCOVA; Time frame: week 12; LSM difference = -1.4, 95% CI 2-sided [-3.0 to 0.2], Standard Error of Mean 0.8
Statistical Analysis 8: Comparison: Placebo vs Gabapentin Enacarbil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.312, ANCOVA; Time frame: EoT; LSM difference = -0.8, 95% CI 2-sided [-2.4 to 0.8], Standard Error of Mean 0.8

3. Secondary Outcome: Percentage of Participants With an Investigator-rated Clinical Global Impression (ICGI) Response
Description: ICGI was assessed by 7-point ordinate scale. Participants who were "Very much improved" or "Much improved" were defined as responders.
Time Frame: EoT (week 12)
Population: FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 188
percentage of participants | 53.2 [45.8 to 60.6] | 57.4 [50.0 to 64.6]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin Enacarbil; Test type: Superiority; p = 0.467, Fisher Exact; difference = 4.2, 95% CI 2-sided [-6.4 to 14.8]

4. Secondary Outcome: Percentage of Participants With a Patient-rated Clinical Global Impression (PCGI) Response
Description: PCGI was assessed by 7-point ordinate scale. Participants who were "Very much improved" or "Much improved" were defined as responders.
Time Frame: EoT (week 12)
Population: FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 188
percentage of participants | 50.5 [43.1 to 57.9] | 56.4 [49.0 to 63.6]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin Enacarbil; Test type: Superiority; p = 0.300, Fisher Exact; difference = 5.8, 95% CI 2-sided [-4.8 to 16.5]

5. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index Total Score (PSQI)
Description: The self-rated items of the PSQI generate seven component scores (range of subscale scores, 0-3). The sum of these seven component scores yielded one global score of subjective sleep quality (range, 0-21). Higher scores represent poorer subjective sleep. ANCOVA model with the baseline value as a covariate was used.
Time Frame: Baseline and EoT (week 12)
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 185 | 187
units on a scale | -1.7 [-2.1 to -1.4] | -1.7 [-2.1 to -1.4]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin Enacarbil; LMS difference (gabapentin enacarbil group minus placebo group) of the changes in PSQI component and global scores from baseline was calculated by visit, using the ANCOVA model with the baseline value as a covariate; Test type: Superiority; p = 0.877, ANCOVA; LSM difference = -0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.3

6. Secondary Outcome: Change From Baseline in Athens Insomnia Scale
Description: Athens Insomnia Scale consisted of 8-item scale (range of subscale scores, 0-3). The scale range of Athens Insomnia was 0-24. Higher scores represent poorer sleep quality. ANCOVA model with the baseline value as a covariate was used.
Time Frame: Baseline and EoT (week 12)
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 187
units on a scale | -2.5 [-2.9 to -2.0] | -2.5 [-2.9 to -2.0]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin Enacarbil; LSM difference (gabapentin enacarbil group minus placebo group) of the changes in total score of Athens insomnia scale from baseline was calculated by visit, using the ANCOVA model with the baseline value as a covariate; Test type: Superiority; p = 0.975, ANCOVA; LSM difference = 0.0, 95% CI 2-sided [-0.7 to 0.7], Standard Error of Mean 0.3

7. Secondary Outcome: Change From Baseline in Restless Legs Syndrome (RLS) Pain Score
Description: The scale range of RLS pain score was 0-10. Higher scores represent greater RLS pain intensity. ANCOVA model with the baseline value as a covariate was used.
Time Frame: Baseline and EoT (week 12)
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 188
units on a scale | -0.9 [-1.2 to -0.7] | -1.0 [-1.2 to -0.7]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin Enacarbil; LSM difference (gabapentin enacarbil group minus placebo group) of the changes in RLS pain score from baseline was calculated by visit, using the ANCOVA model with the baseline value as a covariate; Test type: Superiority; p = 0.838, ANCOVA; LSM difference = -0.0, 95% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.2

8. Secondary Outcome: Change From Baseline in Health Status Score of EuroQol-5 Dimension-5 Level (EQ-5D-5L)
Description: Health status was assessed by general visual analog scale (VAS). The VAS ranges from 0 (worst health status) and 100 (best health status).
Time Frame: Baseline and EoT (week 12)
Population: FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 187
units on a scale | 2.7 (16.7) | 4.2 (15.3)

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events (TEAE) was defined as an adverse event (AE) with onset after the start of the run-in period. A drug-related TEAE was a TEAE with at least a possible relationship to the study drug as assessed by the investigator. Serious TEAE was an AE considered serious.
Time Frame: From first dose of study drug up to week 13
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gabapentin Enacarbil
Number analyzed (Participants) | 186 | 189
Participants
  Any TEAEs | 71 | 94
  Drug-related TEAEs | 36 | 60
  TEAEs leading to death | 0 | 0
  Serious TEAEs | 0 | 3
  Drug-related serious TEAEs | 0 | 0
  TEAEs leading to discontinuation of study drug | 4 | 4
  Drug-related TEAEs leading to disc. of study drug | 3 | 4

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to week 13
Arm/Group | Placebo | Gabapentin Enacarbil
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/189
Serious Adverse Events (participants affected / at risk) | 0/186 | 3/189
Other Adverse Events (participants affected / at risk) | 32/186 | 59/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=186) | Gabapentin Enacarbil (N=189)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=186) | Gabapentin Enacarbil (N=189)
Nasopharyngitis (Infections and infestations) | 20 (22) | 24 (26)
Somnolence neonatal (Nervous system disorders) | 13 (13) | 25 (26)
Dizziness (Nervous system disorders) | 0 (0) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT03053427/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT03053427/SAP_001.pdf